CLINICAL TRIAL: NCT01641406
Title: "Phase II Study of PET Guided Neoadjuvant Chemotherapy (NAC) and Oncotype Guided Hormonal Therapy of Breast Cancer"
Acronym: NACprotocol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Responsible Party: Principal Investigator, Fernando Cabanillas, Hematolgist-Oncologist, Auxilio Mutuo Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC CCAM 11-01; NCT01330212 (obsolete NCT alias)
Record Dates: First submitted 2012-07-11; First posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Infiltrating Duct and Lobular Carcinoma In Situ; Invasive Lobular Breast Carcinoma; Inflammatory Breast Carcinoma
Keywords: NAC Protocol; NAC and Oncotype Guided Hormonal therapy for breast cancer; Neoadjuvant and Oncotype; NAC CCAM 1101
MeSH Terms: conditions — Breast Carcinoma In Situ; Carcinoma, Lobular; Inflammatory Breast Neoplasms | interventions — Docetaxel; Epirubicin; Cyclophosphamide; Vinorelbine; Capecitabine; Trastuzumab; Bevacizumab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ER- (Triple Neg. and ER- PR+ Her 2 -) (Experimental): Experimental chemotherapy using neoadjuvant approach
  Interventions: Drug: Docetaxel, Epirubicin, Cyclophosphamide/Navelbine, Capecitabine, Trastuzumab, Bevacizumab
- Her 2 + (Experimental): Experimental chemotherapy using neoadjuvant approach
  Interventions: Drug: Docetaxel, Epirubicin, Cyclophosphamide/Navelbine, Capecitabine, Trastuzumab, Bevacizumab
- ER + (ER+ PR+ Her 2- / ER+ PR- Her 2 -) (Experimental): Experimental chemotherapy using neoadjuvant approach
  Interventions: Drug: Docetaxel, Epirubicin, Cyclophosphamide/Navelbine, Capecitabine, Trastuzumab, Bevacizumab

INTERVENTIONS:
Drug: Docetaxel, Epirubicin, Cyclophosphamide/Navelbine, Capecitabine, Trastuzumab, Bevacizumab — ER-(Triple Negative and ER-PR+Her-2-):Patients who respond to the first 4 courses of TEC with a Complete Remission will receive 4 more courses of TEC. Patients who respond to the first 4 courses of TEC with a Partial Remission or Stable Disease will then have their treatment changed to the non-cross resistant NAX regimen.Courses will be repeated every 21 days according to blood counts.A total of 4 courses will be given.
  Other Names: Neoadjuvant chemotherapy for breast cancer
  Arms: ER- (Triple Neg. and ER- PR+ Her 2 -)
Drug: Docetaxel, Epirubicin, Cyclophosphamide/Navelbine, Capecitabine, Trastuzumab, Bevacizumab — Her-2 positive cases:Patients who respond to 4 courses of TEC with either a partial or complete remission will then receive 4 additional courses of Docetaxel plus Herceptin, and upon completion of the 4th course of DH they will undergo definitive surgery.A total of 4 courses will be given. Courses will be repeated every 21 days according to blood counts. Patients whose response after 4 courses of TEC is either stable disease or progression, will be treated with "NTX".
  Other Names: Neoadjuvant chemotherapy for breast cancer
  Arms: Her 2 +
Drug: Docetaxel, Epirubicin, Cyclophosphamide/Navelbine, Capecitabine, Trastuzumab, Bevacizumab — ER+ Cases(ER+PR+Her-2- and ER+PR-Her-2-):After the first course of TEC if the SUV of the primary tumor is >5%, treatment will be TEC x 4 courses. If the Oncotype is low, patients will be switched to hormonal therapy x 6 months. If the Oncotype result is intermediate/high, patients will be NAX chemotherapy x 4 courses. If the SUV post course #1 TEC is <5%, subsequent treatment will depend on the Oncotype.If the Oncotype is low, the treatment will be hormonal therapy x 6 months. If the Oncotype is intermediate/high , the treatment will be NAX chemotherapy x 4. Surgery will be performed 6 weeks after the 4th course of NAX chemotherapy.
  Other Names: Neoadjuvant chemotherapy for breast cancer
  Arms: ER + (ER+ PR+ Her 2- / ER+ PR- Her 2 -)

SUMMARY:
The purpose of this study is to evaluate a novel neoadjuvant regimen for invasive breast carcinoma by using the MD Anderson residual cancer burden score.To prospectively evaluate the utility of the PET scan to guide the neoadjuvant treatment and the utility of the Oncotype test as a stratifier for treatment decisons in ER+/Her2- patients. To evaluate the clinical anti-tumor activity of neoadjuvant hormonal therapy in ER+/Her2 negative patients. To evaluate the prognostic factors associated associated with pathological response as measured by the residual cancer burden tool.

DETAILED DESCRIPTION:
Treatment propose of TEC-NAX for the triple negatives and for the Her2+ cases. For the Er+/Her2- cases, we propose to use the PET scan to guide therapy after the first course of TEC. Those who drop in SUV≤5%, will have their treatment modified by using the Oncotype test. Those Her2 negative patients whose response to the first 4 courses of induction TEC is less than a complete remission, will have their tretment changed to a second line regimen, Navelbine-Avastin-Xeloda(NAX), with the intention of capturing a better response prior to surgery. Those who are Her2+ will initially also receive TEC but subsequent therapy will include Trastuzumab(Herceptin) whether thet respond wellor not to TEC.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated (no chemotherapy, hormonal or radiation therapy)invasive breast cancer.
* Diagnosis of invasive ductal or lobular breast cancer plus or minus DCIS. Inflammatory carcinoma will also be elegible.
* Age≥ 18 years
* Only female patients are eligible
* Tumor≥ 1.0cm by MRI and/or sonographic or clinical exam measurements. If the tumor is <1.0 but the patient has biopsy proven lymph node metastasis, she will also be considered eligible.Although only tumors≥2cm are consideredmeasurable by RECIST criteria, we will nevertheless include tumors≥1cm since the primary endpoint is pathological CR rate.
* Performance status ECOG≤2 or Karnofsky≥ 50%
* Peripheral neuropathy≤ grade 1
* Hematologic (minimal values):Absolute Neutrophil count≥1,500/mm³; Hemoglobin≥8.0g/dl; Paltelet count≥100,000/mm³
* Hepatic; Total bilirubin≤ULN AST and ALT and ALP do not have to be within the range. In determining eligibility the more abnormal of the two values(AST or ALT) should be use as per protocol table on p.24of 69.
* Women of childbearing potential must have a negative pregnancy test
* Men and women of childbearing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months thereafter.
* Renal;urine protein:creatinine(UPC)ratio1.0 at screening or urine dipstick for proteinuria<2+(patients discovered to have˃/=2+ protinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate</=1g of protein in 24 hrs to be elegible

Exclusion Criteria:

* Pregnant or breast feeding patients are excluded
* Patients with second malignancies with expected survival<5 years
* Previous chemotherapy with Taxanes,Anthracyclines or Cyclophosphamide.
* Patientes with history of severe hypersensitivity reaction to Taxotere(Docetaxel)or other drugs formulated with polysorbate 80.
* Pure DCIS diagnoses are not elegible
* Special histologies with favorable prognosis such as mucinous, tubular are not elegible
* Patients with reduced ejection fraction<50% are not eligible
* Patients with tumors<1.0cm unless biopsy proven axillary node metastasis present.
* Cardiac thrombotic events in the past 12 months
* Stroke or transient ischemic attacks (TIA) within 12 months
* poorly controlled hypertension defined as persistent blood pressure elevation˃150 systolic and/or 100 diastolic not responsive to medications.
* GI condition that increases risk of perforation within 6 months of study
* Any serious non-healing wound, ulcer, or bone fracture.
* No minor surgical procedure within 7 days of study entry or major surgery within 28 days of study entry or anticipation of need for major surgical procedure during the course of the study.
* Significant vascular disease such as symptomatic peripheral vascular disease.
* Any evidence of bleeding diathesis or coagulopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to obtain a RCB rate of 0-1 in at least 66% | 2 years
  The primary objective is to raise the RCB rate of 0-1 to ≥40%. the startegy of using Oncotype test to guide NAC therapy will be considered encouraging for future testing if we are able to achieve this goal.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — Auxilio Mutuo Hospital Cancer Center
Locations (1):
- Hospital Auxilio Mutuo Cancer Center, San Juan, PR, Puerto Rico